CLINICAL TRIAL: NCT00279175
Title: Reinfusion of Enriched Progenitor Cells And Infarct Remodeling in Acute Myocardial Infarction (REPAIR - AMI)
Brief Title: REPAIR-AMI: Intracoronary Progenitor Cells in Acute Myocardial Infarction (AMI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A. M. Zeiher (Other)
Collaborators: Johann Wolfgang Goethe University Hospital (Other); Blutspendedienst Baden-Württemberg - Hessen (Unknown); Guidant Corporation (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, A. M. Zeiher, Professor Dr. med., Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2/04; Paul-Ehrlich-Institute 1034/01; EudraCT 2006-000250-43
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Myocardial Infarction
Keywords: Acute myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- BMC (Experimental): Intracoronary infusion of autologous bone marrow derived cells
  Interventions: Biological: Intracoronary infusion of enriched bone marrow-derived progenitor cells
- Placebo (Placebo Comparator): Intracoronary infusion of Placebo medium
  Interventions: Biological: Placebo medium supplemented with autologous serum

INTERVENTIONS:
Biological: Intracoronary infusion of enriched bone marrow-derived progenitor cells
  Arms: BMC
Biological: Placebo medium supplemented with autologous serum
  Arms: Placebo

SUMMARY:
Impaired contractile function after a heart attack of the heart is a major cause of "heart failure" limiting quality of life and prognosis, which cannot be prevented even with optimal standard therapy, including immediate balloon/stent dilation of the infarct vessel.

The aim of the REPAIR-AMI trial is to investigate whether infusion of progenitor cells into the infarct vessel (after successful reperfusion therapy) may improve left ventricular contractile function compared to placebo therapy. After bone marrow aspiration progenitor cells are enriched via a centrifugation method.

DETAILED DESCRIPTION:
* The study is a double-blind, placebo-controlled, randomized, multicenter trial.
* Patients after an acute myocardial infarction, undergoing successful reperfusion therapy are included.
* All patients undergo bone marrow aspiration 3 to 6 days after the infarction.
* After cell processing, enriched bone marrow-derived progenitor cells or placebo medium is infused direct into the infarct related artery during stop-flow. In addition, a left ventricular angiography is performed.
* After 4 months left ventricular angiography is repeated. The primary endpoint is the difference in change of left ventricular ejection fraction between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myocardial infarction (ST elevation in at least 2 leads >= 0.2 mV in V1,V2 or V3 or >= 0.1 mV in other leads), treated by one of the following procedures

  * Either acute PCI with stent implantation within 24 hours after symptom onset or
  * treatment with thrombolysis within 12 hours of symptom onset followed by PCI with stent implantation within 24 hours after thrombolysis.
* Acute PCI / stent implantation has been successful (residual stenosis visually < 30% and TIMI flow >= 2).
* At the time of inclusion patient does no longer require i.v. catecholamines or mechanical hemodynamic support (aortic balloon pump)
* Significant regional wall motion abnormality in LV angiogram at the time of acute PCI (ejection fraction <= 45% on visual estimation).
* Maximal CK elevation >= 400 U/l (measured at 37° C) with significant MB fraction > 6%
* Age 18 - 80 Years
* Written informed consent

Exclusion Criteria:

* Regional wall motion abnormality outside the area involved in the index acute myocardial infarction.
* Need to revascularize additional vessels, outside the infarct artery.
* Arteriovenous malformations or aneurysms
* Active infection (CRP > 10 mg/dl) now, or fever or diarrhea within last 4 weeks.
* Chronic inflammatory disease
* HIV infection or active hepatitis
* Neoplastic disease without documented remission within the past 5 years.
* Cerebrovascular insult within 3 months
* Impaired renal function (creatinine > 2 mg/dl) at the time of cell therapy
* Significant liver disease (GOT > 2x upper limit) or spontaneous INR > 1,5)
* Anemia (hemoglobin < 8.5 mg/dl)
* Platelet count < 100.000/µl
* Hypersplenism
* Known allergy or intolerance to clopidogrel, heparin or abciximab.
* History of bleeding disorder
* Gastrointestinal bleeding within 3 months
* Major surgical procedure or traumata within 2 months
* Uncontrolled hypertension
* Pregnancy
* Mental retardation
* Previously performed stem / progenitor cell therapy
* Participation in another clinical trial within the last 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2004-04; Primary Completion 2005-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in global left ventricular function in quantitative LV angiography after 4 months. | baseline to 4 months
  absolute delta LVEF (%)

SECONDARY OUTCOMES:
Primary endpoint in patients without restenosis. | baseline to 4 months
  absolute delta LVEF (%)
Improvement of regional wall motion in infarct area | baseline to 4 months
Reduction of LV end-systolic volume | baseline to 4 months
Major adverse cardiac events (MACE) | at 4, 12 and 60 months
Rehospitalization due to heart failure. | 4, 12, 60 months
NYHA status after 12 months | 12 months
Amendment for extended follow up after 2 and 5 years: | 24 and 60 months
outcomes in major adverse cardiac events (MACE) | 4, 12, 60 months
Rehospitalization due to heart failure | 4, 12, 60 months
NYHA status | 4, 12, 60 months
patients in MRI subgroup: improvement in left ventricular function | 4, 12, 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Zeiher, MD, Principal Investigator — J. W. Goethe University Hospitals; Volker Schächinger, MD, Study Director — J. W. Goethe University Hopspitals
Locations (17):
- Germany (16):
  - Zentralklinik Bad Berka, Bad Berka
  - Kerckhoff Klinik, Bad Nauheim
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - BG Kliniken Bergmannsheil, Bochum
  - Klinikum Lippe, Detmold
  - Rotes-Kreuz Krankenhaus - Kardiologisches Centrum, Frankfurt
  - J. W. Goethe University Hospitals, Frankfurt
  - Universitätsklinkum Giessen, Giessen
  - Parxis Schofer, Mathey und Partner, Hamburg
  - Universitätsklikum Homburg, Homburg/Saar
  - Klinikum Kassel, Kassel
  - Herzzentrum - Universität Leipzig, Leipzig
  - Herzzentrum Ludwigshafen, Ludwigshafen
  - Universitätsklinik Mainz, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - Zentralklinikum Suhl, Suhl
- Universitätsspital Zürich, Zurich, Switzerland

REFERENCES:
- [Background] Schachinger V, Tonn T, Dimmeler S, Zeiher AM. Bone-marrow-derived progenitor cell therapy in need of proof of concept: design of the REPAIR-AMI trial. Nat Clin Pract Cardiovasc Med. 2006 Mar;3 Suppl 1:S23-8. doi: 10.1038/ncpcardio0441. PMID 16501626
- [Result] Schachinger V, Erbs S, Elsasser A, Haberbosch W, Hambrecht R, Holschermann H, Yu J, Corti R, Mathey DG, Hamm CW, Suselbeck T, Assmus B, Tonn T, Dimmeler S, Zeiher AM; REPAIR-AMI Investigators. Intracoronary bone marrow-derived progenitor cells in acute myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1210-21. doi: 10.1056/NEJMoa060186. PMID 16990384
- [Result] Schachinger V, Erbs S, Elsasser A, Haberbosch W, Hambrecht R, Holschermann H, Yu J, Corti R, Mathey DG, Hamm CW, Suselbeck T, Werner N, Haase J, Neuzner J, Germing A, Mark B, Assmus B, Tonn T, Dimmeler S, Zeiher AM; REPAIR-AMI Investigators. Improved clinical outcome after intracoronary administration of bone-marrow-derived progenitor cells in acute myocardial infarction: final 1-year results of the REPAIR-AMI trial. Eur Heart J. 2006 Dec;27(23):2775-83. doi: 10.1093/eurheartj/ehl388. Epub 2006 Nov 10. PMID 17098754
- [Result] Dill T, Schachinger V, Rolf A, Mollmann S, Thiele H, Tillmanns H, Assmus B, Dimmeler S, Zeiher AM, Hamm C. Intracoronary administration of bone marrow-derived progenitor cells improves left ventricular function in patients at risk for adverse remodeling after acute ST-segment elevation myocardial infarction: results of the Reinfusion of Enriched Progenitor cells And Infarct Remodeling in Acute Myocardial Infarction study (REPAIR-AMI) cardiac magnetic resonance imaging substudy. Am Heart J. 2009 Mar;157(3):541-7. doi: 10.1016/j.ahj.2008.11.011. Epub 2009 Jan 31. PMID 19249426
- [Result] Erbs S, Linke A, Schachinger V, Assmus B, Thiele H, Diederich KW, Hoffmann C, Dimmeler S, Tonn T, Hambrecht R, Zeiher AM, Schuler G. Restoration of microvascular function in the infarct-related artery by intracoronary transplantation of bone marrow progenitor cells in patients with acute myocardial infarction: the Doppler Substudy of the Reinfusion of Enriched Progenitor Cells and Infarct Remodeling in Acute Myocardial Infarction (REPAIR-AMI) trial. Circulation. 2007 Jul 24;116(4):366-74. doi: 10.1161/CIRCULATIONAHA.106.671545. Epub 2007 Jul 9. PMID 17620510
- [Result] Assmus B, Rolf A, Erbs S, Elsasser A, Haberbosch W, Hambrecht R, Tillmanns H, Yu J, Corti R, Mathey DG, Hamm CW, Suselbeck T, Tonn T, Dimmeler S, Dill T, Zeiher AM, Schachinger V; REPAIR-AMI Investigators. Clinical outcome 2 years after intracoronary administration of bone marrow-derived progenitor cells in acute myocardial infarction. Circ Heart Fail. 2010 Jan;3(1):89-96. doi: 10.1161/CIRCHEARTFAILURE.108.843243. Epub 2009 Dec 8. PMID 19996415
- [Derived] Rolf A, Assmus B, Schachinger V, Rixe J, Mollmann S, Mollmann H, Dimmeler S, Zeiher AM, Hamm CW, Dill T. Maladaptive hypertrophy after acute myocardial infarction positive effect of bone marrow-derived stem cell therapy on regional remodeling measured by cardiac MRI. Clin Res Cardiol. 2011 Nov;100(11):983-92. doi: 10.1007/s00392-011-0330-3. Epub 2011 Jun 17. PMID 21681619
- [Derived] Assmus B, Tonn T, Seeger FH, Yoon CH, Leistner D, Klotsche J, Schachinger V, Seifried E, Zeiher AM, Dimmeler S. Red blood cell contamination of the final cell product impairs the efficacy of autologous bone marrow mononuclear cell therapy. J Am Coll Cardiol. 2010 Mar 30;55(13):1385-94. doi: 10.1016/j.jacc.2009.10.059. PMID 20338501